CLINICAL TRIAL: NCT06277076
Title: Accuracy of Computer- Guided Implant Surgery in Partially Edentulous Patients: a Prospective Observational Study.
Brief Title: Accuracy of Computer- Guided Implant Surgery in Partially Edentulous Patients.
Status: Completed | Type: Observational
Sponsor: Saint-Joseph University (Other)
Responsible Party: Principal Investigator, Emile Chrabieh, Principal investigator, Head of Implant Dentistry Diploma program, Clinical Adjunct Professor., Saint-Joseph University
Other Study IDs: FMD1234
Record Dates: First submitted 2024-01-13; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Dental Implant; Computer
Keywords: dental implant; Accuracy; Computer-aided design (CAD); Guided surgery; Surgical guide; Surgical template; Computer-aided manufacturing (CAM)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Computer Implant guided Surgery — Dental implant placed using printed guide after a digital planification on a superimposed 3D surface scan and a 3D Cone Beam imaging of the jaw.

SUMMARY:
The dental implant placed freehand with a digital planing is vastly increasing. The accuracy between the planned and the placed implants still not well determined. Between a single implant and a full mouth rehabilitation, the precision is very wide. A precision scale must be settled according to each indication in order to offer the clinician a safety and a predictability for his procedures.

DETAILED DESCRIPTION:
In this paper the investigators report an original research evaluating the accuracy of computer-guided implant placement in posterior edentulous mandibular spaces. In this randomized controlled trial, several factors were evaluated such as primary implant stability, possibility of immediate loading, displacement at crestal and apical levels, angle of deviation, surgical guide design, computer-aided design and computer-aided manufacturing accuracy, and variance between different implant macro-geometries and lengths. As exhaustive description of the assessment techniques as well as the statistic results were also presented in this article.

Nowadays, the use of guided surgery is vastly increasing in a daily dental practice. In the "Era of Digital Dentistry", it is of utmost importance to evaluate the accuracy and precision of the computer-guided techniques in order to determine their limits, avoid risks (adjacent anatomical structures, limited crestal volume, immediate loading), and apply them in safe manner. Evidence-based scientific data on this matter is still deficient. In these terms, the investigators consider it very interesting and of high clinical value for all oral surgeons and dental practitioners to evaluate in a clinical research the precision and distortion of computer-guided implant surgery.

ELIGIBILITY:
Inclusion Criteria:

* Acceptable oral hygiene with no signs of active periodontal disease or local infection
* American Society of Anesthesiologists (ASA) physical status classification 1 and 2
* Non or Light smoking (< 10 cigarettes per day)
* Acceptable intermaxillary space (44 mm minimum)
* Minimal crestal width of 5.5mm
* Minimal residual bone height of 10mm above the alveolar nerve canal

Exclusion Criteria:

* Head and neck irradiation
* Bone grafted sites
* Severe bruxism
* Cone Beam Computed tomography with exaggerated artifacts
* Limited intermaxillary space

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients presenting at Saint Joseph University of Beirut dental clinics with a distal-shortened mandible or distal intercalary space of two to three missing premolars or molars (class I, II or VI according to Kennedy's classification on edentulous spaces) and requiring implant-supported reconstructions were selected to participate in this study.
  For each case two implants were placed with a fully guided procedure. Thirteen patients were included in this study with twenty-five implants eligible for accuracy evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2023-01-28 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Assess Accuracy of Implant Placement in Vertical Displacement (VD). | 4 months
  Evaluate the accuracy of implant placement by comparing the planned positions (from the computer) with the actual positions of the placed implants (using the printed guide). The tool to assess the accuracy/deviation is a software that superimpose two "Digital Imaging and Communications in Medicine" (DCM) Files of the planned and the actual position implants. the first DCM issued from the planning software and second DCM file after scanning the implant in the jaw. The first outcome measure was provided to calculate the amount of distortion in millimeter (mm) for the Vertical Displacement (VD) (mm).
Assess Accuracy of Implant Placement in Horizontal Displacement (HD) | 4 months
  Evaluate the accuracy of implant placement by comparing the planned positions (from the computer) with the actual positions of the placed implants (using the printed guide). The tool to assess the accuracy/deviation is a software that superimpose two "Digital Imaging and Communications in Medicine" (DCM) Files of the planned and the actual position implants. the first DCM issued from the planning software and second DCM file after scanning the implant in the jaw. The second outcome measure was provided to calculate the amount of distortion in millimeter (mm) for the Horizontal Displacement (HD).
Assess Accuracy of Implant Placement in Error Depth (ED) | 4 months
  Evaluate the accuracy of implant placement by comparing the planned positions (from the computer) with the actual positions of the placed implants (using the printed guide). The tool to assess the accuracy/deviation is a software that superimpose two "Digital Imaging and Communications in Medicine" (DCM) Files of the planned and the actual position implants. the first DCM issued from the planning software and second DCM file after scanning the implant in the jaw. The third outcome measure was provided to calculate the amount of distortion in millimeter (mm) for the Error Depth (ED) (mm).
Assess Accuracy of Implant Placement in Error Angle (EA) | 4 months
  Evaluate the accuracy of implant placement by comparing the planned positions (from the computer) with the actual positions of the placed implants (using the printed guide). The tool to assess the accuracy/deviation is a software that superimpose two "Digital Imaging and Communications in Medicine" (DCM) Files of the planned and the actual position implants. the first DCM issued from the planning software and second DCM file after scanning the implant in the jaw. The fourth outcome measure was provided to calculate the amount of distortion in in degree of the Error Angle (EA).

SECONDARY OUTCOMES:
Evaluate Precision of the Printed Guide | 4 months
  Assess how precisely the printed guide translates the planned positions to the actual implant placements. Using the same assessment tool as for the primary outcome measure.
Study Complications and Adverse Events | 4 months
  Monitor and report any complications or adverse events associated with the use of the printed guide during implant placement.

CONTACTS AND LOCATIONS:
Overall Officials: Emile Chrabieh, Master, Principal Investigator — Faculty at the dental school, oral surgery department, Saint Joseph University of Beirut
Locations (1):
- Saint Joseph University of Beirut/Dental school, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Younes F, Cosyn J, De Bruyckere T, Cleymaet R, Bouckaert E, Eghbali A. A randomized controlled study on the accuracy of free-handed, pilot-drill guided and fully guided implant surgery in partially edentulous patients. J Clin Periodontol. 2018 Jun;45(6):721-732. doi: 10.1111/jcpe.12897. Epub 2018 May 10. PMID 29608793
- [Background] Li J, Chen Z, Chan HL, Sinjab K, Yu H, Wang HL. Does flap opening or not influence the accuracy of semi-guided implant placement in partially edentulous sites? Clin Implant Dent Relat Res. 2019 Dec;21(6):1253-1261. doi: 10.1111/cid.12847. Epub 2019 Oct 23. PMID 31642588
- [Background] Arisan V, Karabuda CZ, Ozdemir T. Implant surgery using bone- and mucosa-supported stereolithographic guides in totally edentulous jaws: surgical and post-operative outcomes of computer-aided vs. standard techniques. Clin Oral Implants Res. 2010 Sep;21(9):980-8. doi: 10.1111/j.1600-0501.2010.01957.x. Epub 2010 May 24. PMID 20497439
- [Background] van Steenberghe D, Molly L, Jacobs R, Vandekerckhove B, Quirynen M, Naert I. The immediate rehabilitation by means of a ready-made final fixed prosthesis in the edentulous mandible: a 1-year follow-up study on 50 consecutive patients. Clin Oral Implants Res. 2004 Jun;15(3):360-5. doi: 10.1111/j.1600-0501.2004.01069.x. PMID 15142100
- [Background] Tahmaseb A, Wu V, Wismeijer D, Coucke W, Evans C. The accuracy of static computer-aided implant surgery: A systematic review and meta-analysis. Clin Oral Implants Res. 2018 Oct;29 Suppl 16:416-435. doi: 10.1111/clr.13346. PMID 30328191